CLINICAL TRIAL: NCT01109680
Title: A Single Center, Open-Label Study to Quantify Metabolites of [14C]-Neramexane in Plasma and Urine in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Dr. Dirk Garmann, Merz Pharmaceuticals GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MRZ 92579-1048-0
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2010-04

CONDITIONS: Metabolism of Neramexane
MeSH Terms: interventions — neramexane

ARMS (1):
- 14 C labelled Neramexane, capsule (Experimental)
  Interventions: Drug: Neramexane

INTERVENTIONS:
Drug: Neramexane — Multiple dose Neramexane followed by single dose 14C Neramexane

SUMMARY:
A Single Center, Open-Label Study to quantify metabolites of [14C]-Neramexane in plasma and urine in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 to 65 years inclusive
* BMI of 18-29 kg/m2 (inclusive) and a body weight of ≥50 and ≤90 kg
* All ethnicities, Fitzpatrick type < IV (see appendix 2)
* Willing and able to provide written informed consent after having been informed of the requirements and the restrictions of the study
* Healthy adult male subject, who is able to read, to write and fully understand Dutch language

Exclusion Criteria:

* History of clinically relevant allergy or known hypersensitivity to Neramexane/Memantine/Amantadine and their derivates
* Exposure to another investigational agent within the last two months before first drug administration
* Administration of radiolabeled substance or exposure to significant radiation (e.g. serial X-ray or CT scans etc.) within the last 12 months. X-rays or spiral CT scans of extremities are allowed.

Lack of suitability for the study

* Any evidence of a significant cardiovascular, pulmonary, renal, hepatic, gastrointestinal, endocrinological, metabolic, psychiatric, neurologic or other acute or chronic disease
* Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the pharmacokinetics of the investigational medicinal products (e.g. cholecystectomy, active gastric ulcers, etc.)
* Clinically relevant acute or chronic infections, observed within 4 weeks before first drug administration
* History of malignancy, except basal cell carcinoma
* Any clinically relevant deviation in clinical or laboratory assessment as deemed by the investigator
* Abnormalities in the 12-lead ECG (at screening) which in the discretion of the investigator and the Merz scientific expert are clinical relevant or might affect the study objectives
* Systolic blood pressure <95 mmHg or >155 mmHg or diastolic blood pressure < 50 mmHg or >95 mmHg in supine position
* Pulse rate <45 or >100 beats per minute
* History of alcohol or drug dependence
* Alcohol consumption averaging a weekly intake in excess of 21 units of alcohol (one unit of alcohol equals a glass of beer of 300 mL, a glass of wine of 125 mL, or a measure of spirits of 25 mL) within the last year
* Regular large caffeine consumption averaging more than 6 cups of coffee and/or tea per day or more than 1 L of caffeine-containing beverages per day within the last year
* Use of any prescribed medication 4 weeks prior to the first administration of IMP (except paracetamol, maximum 2 g/day). Thyroid hormone substitution will be allowed)
* Regular use of over-the-counter drugs 4 weeks prior to the first administration of the IMP.
* Occasional use of OTC drugs (except paracetamol, maximum 2 g/day) in the 2 weeks prior to the first administration of the IMP
* Use of any food, food supplement or medication known to induce or inhibit CYP3A4 or other cytochrome P450 enzymes within two weeks before first drug administration e.g. grapefruit, St. Johns wort
* Consume of xanthine derivates (including caffeine) within two days before first drug administration
* Smokers or ex-smokers who have stopped for less than 6 months, and user of snuff, nicotine replacement chewing tobacco
* Blood donation more than 450 mL within 60 days before first drug administration
* Positive results in any of the serology tests
* Positive drug screen or alcohol test
* Subject is an employee or direct relative of an employee of the CRO or Merz Pharmaceuticals
* Lack of ability or willingness to give informed consent
* Lack of willingness or inability to co-operate adequately
* Vulnerable subjects (e.g. persons kept in detention)
* Anticipated non-availability for study visits/procedures

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Metabolite Profiling

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services, Antwerp, Belgium